CLINICAL TRIAL: NCT06157684
Title: Assessment of the Effect of Postprandial Ambulation on Birth Weight Percentile in Patients With Gestational Diabetes Mellitus.
Brief Title: Timing of Ambulation and Infant Birth Weight in Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Anna Whelan, Clinical and Research Fellow, Principal Investigator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDMAmbulation_WIH
Record Dates: First submitted 2023-04-20; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Gestational Diabetes; Pregnancy Complications; Pregnancy in Diabetic; Fetal Macrosomia
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy Complications; Pregnancy in Diabetics; Fetal Macrosomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postprandial Ambulation (Experimental): Participants are counseled to walk for 20 minutes within 2 hours following meals daily.
  Interventions: Behavioral: Postprandial ambulation
- Routine exercise counseling (No Intervention): Participants are counseled on routine ADA recommendations for 30 minutes of low-impact exercise 5 times a week

INTERVENTIONS:
Behavioral: Postprandial ambulation — See arm description
  Arms: Postprandial Ambulation

SUMMARY:
This is a randomized controlled trial to assess the effect of routine exercise counseling compared to the recommendation for postprandial ambulation on infant birthweight among pregnant people with gestational diabetes mellitus.

The primary outcome is birthweight percentile for gestational age at delivery.

Secondary outcomes include feasibility and acceptability, need for metformin or insulin for glycemic control, mode of delivery, neonatal hypoglycemia.

Participants will be counseled to either complete 20 minutes of walking after meals, or be counseled with routine exercise counseling of 30 minutes of low-impact 5x a week. Their activity will be tracked by "FitBit" pedometers and uploaded via bluetooth to a database for review. They will continue to receive routine obstetric and diabetes care.

DETAILED DESCRIPTION:
This is a randomized controlled trial of postprandial ambulation to decrease birthweight percentile in patients with gestational diabetes.

Patients who are diagnosed with gestational diabetes. and enrolled in the Diabetes in Pregnancy Program in the Division of Maternal Fetal Medicine at Women and Infants Hospital of Rhode Island will be approach for inclusion in the study. After consent is obtained, patients with gestational diabetes. will be randomized into one of two groups.

* Group 1: intervention group: 20 minutes of walking after meals
* Group 2: non-intervention group: routine activity

Randomization will occur via computer generated randomization in blocks of 10. After consent is obtained the participants will be randomized via REDCap. They will then receive counseling specific to their group. They will be provided with an activity monitor and instructed on how to use as well as charge and upload data. They will be provided with the information from the manufacturer as well as trouble shooting guide.

As is the standard of care in this clinic, both groups would be equipped with glucometers and diabetic testing supplies. Both groups would receive the same diabetes and nutrition counseling from qualified nursing staff. Additionally, all participants will be provided with Bluetooth enabled pedometers. Those participants assigned to the intervention group would be instructed to walk for 20 minutes within the first two hours following each meal, while those assigned to the routine activity group will receive standard exercise counseling per American College of Obstetricians and Gynecologists and the American Diabetes Association.

Patients will touch base weekly (either in person or by email) with diabetic nurse educators as is the standard management in this clinic. The decision to start insulin for glucose management will remain up to the discretion of the participant's medical doctor. In addition to review of their glucose logs, patients will review activity log and pedometer data with research staff on a weekly or biweekly basis.

Delivery data will be collected on all patients including routine postpartum laboratory data.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with gestational diabetes and receive care at the Maternal Fetal Medicine Diabetes in Pregnancy Program and who are fluent in English or Spanish.

Exclusion Criteria:

* Pre-existing type 1 or type 2 diabetes, and those diagnosed with gestational diabetes in the first trimester. Patients who are either physically unable to ambulate or who have other contraindications to ambulation.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Infant birthweight percentile | Single time point - at birth
  Birthweight percentile for gestational age for neonatal sex

SECONDARY OUTCOMES:
infant birthweight | Single time point - at birth
  birthweight measured after delivery
neonatal hypoglycemia treatment | within 48 hours of birth
  need for PO or IV treatment for neonatal hypoglycemia
mode of delivery | Single time point
  spontaneous vaginal, operative vaginal, cesarean delivery
fetal macrosomia | Single time point - at birth
  birthweight >4500 gm
need for insulin or metformin during pregnancy | from diagnosis to delivery of infant
  need for initiation of anti-hyperglycemic treatment during pregnancy

OTHER OUTCOMES:
feasibility and acceptability | 3 months after the study conclusion
  Likert scale for participant experience

CONTACTS AND LOCATIONS:
Locations (1):
- Women & Infants Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT06157684/Prot_000.pdf
  • Informed Consent Form (2022-03-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT06157684/ICF_001.pdf